CLINICAL TRIAL: NCT01398982
Title: The Use of Transversus Abdominis Plane (TAP) Block in Autologous Breast Reconstruction Donor Site: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: TAP Block in DIEP or Free MS-TRAM Donor Site: A RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Society of Plastic Surgeons (Other); The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0969-A
Record Dates: First submitted 2011-07-18; First posted 2011-07-21 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Transversus Abdominis Plane (TAP) Block Catheter; DIEP or Free MS-TRAM Breast Reconstruction; Local Pain Management; Abdominal/ Donor Site
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotonic saline (control group) (Placebo Comparator): At the conclusion of the surgery, a 0.2 mL/kg bolus of Saline will be injected through each catheter in the OR. At midnight following the OR, 0.2mL/Kg of Saline will be injected through each catheter every 8 hours for the next 2 postoperative days by a MD member of the pain team. At 8am on postoperative day 3, the TAP catheters were removed by the pain team. Our rationale for decreasing the frequency of intermittent boluses from every 12 hours to 8 hours in this study design was based on our finding in the pilot study that patients frequently used more PCA between 8-12 hours following Bupivacaine bolus as the effect of the anaesthetic agent weaned off.
  Interventions: Drug: Isotonic saline (control group)
- Bupivacaine (study group) (Experimental): At the conclusion of the surgery, a 0.2 mL/kg bolus of 0.25% Bupivacaine will be injected through each catheter in the OR. At midnight following the OR, 0.2mL/Kg of 0.25% Bupivacaine will be injected through each catheter every 8 hours for the next 2 postoperative days by a MD member of the pain team. At 8am on postoperative day 3, the TAP catheters were removed by the pain team. Our rationale for decreasing the frequency of intermittent boluses from every 12 hours to 8 hours in this study design was based on our finding in the pilot study that patients frequently used more PCA between 8-12 hours following Bupivacaine bolus as the effect of the anaesthetic agent weaned off.
  Interventions: Drug: Bupivacaine (study group); Drug: Isotonic saline (control group)

INTERVENTIONS:
Drug: Bupivacaine (study group) — At the conclusion of the surgery, a 0.2 mL/kg bolus of 0.25% Bupivacaine will be injected through each catheter in the OR. At midnight following the OR, 0.2mL/Kg of 0.25% Bupivacaine will be injected through each catheter every 8 hours for the next 2 postoperative days by a MD member of the pain team. At 8am on postoperative day 3, the TAP catheters were removed by the pain team. Our rationale for decreasing the frequency of intermittent boluses from every 12 hours to 8 hours in this study design was based on our finding in the pilot study that patients frequently used more PCA between 8-12 hours following Bupivacaine bolus as the effect of the anaesthetic agent weaned off.
  Arms: Bupivacaine (study group)
Drug: Isotonic saline (control group) — At the conclusion of the surgery, a 0.2 mL/kg bolus of Saline will be injected through each catheter in the OR. At midnight following the OR, 0.2mL/Kg of Saline will be injected through each catheter every 8 hours for the next 2 postoperative days by a MD member of the pain team. At 8am on postoperative day 3, the TAP catheters were removed by the pain team. Our rationale for decreasing the frequency of intermittent boluses from every 12 hours to 8 hours in this study design was based on our finding in the pilot study that patients frequently used more PCA between 8-12 hours following Bupivacaine bolus as the effect of the anaesthetic agent weaned off.

SUMMARY:
Breast reconstruction using a patient's own abdominal tissue is one of the most common methods for restoring mastectomy defects for breast cancer patients. Despite its increasing popularity and safety, the abdomen remains a major source of postoperative pain. Adequate pain control is important as it has been shown to reduce medical complications, in-hospital death, shortens hospital stay, lessen chronic pain and disability, and in turn lower health-care costs. The current postoperative pain relief protocol consists primarily of a patient-controlled anesthesia device delivering intravenous opioids. Opioids can cause numerous side-effects such as sedation, headache, nausea, vomiting, breathing difficulties, bladder and bowel dysfunction. A promising approach to provide postoperative pain control of the abdominal incision is the newly developed transversus abdominis plane (TAP) peripheral nerve block. Although the TAP block has been found to be an effective pain-relief following major abdominal surgeries, its use has never been studied for breast reconstruction using abdominal tissue. Therefore, the investigators propose to rigorously study the efficacy of a TAP block in reducing postoperative abdominal pain following abdominal tissue breast reconstruction. This study has significant implications in improving both clinical care and health outcomes in patients undergoing this common method of breast reconstruction technique.

DETAILED DESCRIPTION:
1. Statement of Objectives/Specific Aims

The transversus abdominis plane (TAP) block is a newly developed block involving T6-L1 nerves that supply the anterior abdominal wall. Its effectiveness has been reported following major abdominal surgeries, but not following abdominally-based autologous tissue breast reconstruction. Thus, we propose a randomized, double-blind, placebo-controlled trial to evaluate the efficacy of TAP block in improving pain symptomatology following abdominally-based, autologous tissue breast reconstruction.

The primary objective of this study is to compare the mean total opioid consumption in the first postoperative 48 hours between the control and study groups in intravenous morphine equivalent units. By directly blocking the neural afferents, the mean opioid consumption will be significantly lower in the group receiving intermittent local anaesthetic boluses compared to the placebo group through a TAP catheter.

The secondary outcomes of interest are to compare the following parameters:

A. Continuous outcomes i. Total in-hospital cumulative opioid consumption ii. Total in-hospital cumulative anti-nausea consumption iii. Quality of Recovery (QOR) score (0-18) iv. Duration of hospital stay

B. Repeated measures outcomes

In Hospital postoperative measures:

i. Daily pain intensity scores at rest and with movement using a visual pain analogue scale (0-10) ii. Postoperative nausea and vomiting (score of 0-3) iii. Sedation score

Long-term chronic pain, anxiety, function, and quality of life (QOL) measures:

iv. Pain disability index v. Short-form McGill Pain Questionnaire vi. Hospital Anxiety and Depression Scale vii. Short-form 36

C. Time to event outcomes i. Time to first bowel movement ii. Time to ambulation

Hypothesis: Compared to the control group, the TAP block group will have a statistically significant reduction in total in-hospital consumption of opioids, pain scores and side-effects from opioid use such as sedation, nausea, and vomiting. This should also result in a greater QOR score in the TAP block group. Surgical milestones such as time to ambulation, first bowel movement, and duration of hospital stay will also be reduced in the TAP block group. In addition, we hypothesize less acute postoperative pain achieved using the TAP block will result in a reduction in chronic pain and disability, anxiety and depression, and improved QOL in the long-term.

ELIGIBILITY:
Inclusion Criteria:

-Pre-operative eligibility:

* Patients above the age of 18, no upper age limit
* English-speaking
* Delayed reconstruction (mastectomy already performed) or immediate reconstruction (mastectomy at the same time as reconstruction)
* Reconstruction using abdominal tissues including free MS-TRAM or DIEP

Exclusion Criteria:

* Patient refusal
* Inability to give informed consent
* BMI > 40
* Allergy to Bupivacaine
* Known cardiac or liver disease (contraindicated for Bupivacaine use)
* Patients who will undergo any of the following:

  * Implant breast reconstruction
  * Combined implant and autologous tissue reconstruction
  * Non-abdominally based autologous tissue reconstruction
  * Nonmicrosurgical abdominally based breast reconstruction (pedicled TRAM flap)
* Drug addiction
* Opioid tolerance defined as preoperative opioid use of >50 mg PO morphine equivalent
* Psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Zhong, MD, MHS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Zhong T, Ojha M, Bagher S, Butler K, Srinivas C, McCluskey SA, Clarke H, O'Neill AC, Novak CB, Hofer SOP. Transversus abdominis plane block reduces morphine consumption in the early postoperative period following microsurgical abdominal tissue breast reconstruction: a double-blind, placebo-controlled, randomized trial. Plast Reconstr Surg. 2014 Nov;134(5):870-878. doi: 10.1097/PRS.0000000000000613. PMID 25347623
- [Derived] Zhong T, Ojha M, Bagher S, Butler K, O'Neill AC, McCluskey SA, Clarke H, Hofer SO, Srinivas C. Transversus abdominis plane block following abdominally based breast reconstruction: study protocol for a randomized controlled trial. Trials. 2013 Dec 10;14:424. doi: 10.1186/1745-6215-14-424. PMID 24325953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isotonic Saline (Control Group) | Bupivacaine (Study Group)
Started | 44 | 49
Completed | 38 | 47
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isotonic Saline (Control Group) | Bupivacaine (Study Group) | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (8.4) | 52.1 (8.3) | 51.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 49 | 93
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Opioid Consumption
Description: The primary objective of this study is to compare the mean total opioid consumption in the first postoperative 48 hours between the control and study groups in intravenous morphine equivalent units. By directly blocking the neural afferents, the mean opioid consumption will be significantly lower in the group receiving intermittent local anaesthetic boluses compared to the placebo group through a TAP catheter.
Time Frame: first postoperative 48 hours
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Isotonic Saline (Control Group); Bupivacaine (Study Group): At the conclusion of the surgery, a 0.2 mL/kg bolus of 0.25% Bupivacaine or Saline will be injected through each catheter in the OR. At midnight following the OR, 0.2mL/Kg of 0.25% Bupivacaine or Saline will be injected through each catheter every 8 hours for the next 2 postoperative days by a MD member of the pain team. At 8am on postoperative day 3, the TAP catheters were removed by the pain team. Our rationale for decreasing the frequency of intermittent boluses from every 12 hours to 8 hours in this study design was based on our finding in the pilot study that patients frequently used more PCA between 8-12 hours following Bupivacaine bolus as the effect of the anaesthetic agent weaned off.
Arm/Group | Isotonic Saline (Control Group) | Bupivacaine (Study Group)
Number analyzed (Participants) | 38 | 47
mg | 30.0 (19.1) | 20.7 (20.1)
Statistical Analysis 1: Comparison: Isotonic Saline (Control Group) vs Bupivacaine (Study Group); Test type: Non-Inferiority or Equivalence — Based on our published prospective, nonrandomized study using TAP block in abdominally-based autologous tissue breast reconstruction, 40 patients per group would achieve 85% power to detect a 65% reduction in mean total opioid consumption between the control and study groups (significance level alpha = 0.05; using a two-sided Wilcoxon rank-sum test); p = 0.02, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total In-hospital Cumulative Opioid Consumption
Description: Total in-hospital cumulative opioid consumption levels
Time Frame: In-patient hospital stay average of 4 - 5 days
Reporting Status: Not Posted

3. Secondary Outcome: Daily Pain Intensity Scores at Rest and With Movement
Description: Daily pain intensity scores at rest and with movement using a visual pain analogue scale (0-10)
Time Frame: In Hospital postoperative measures, average 4-5 days
Reporting Status: Not Posted

4. Secondary Outcome: Pain Disability
Description: Pain Disability Index Scores
Time Frame: Hospital discharge, average 4-5 days, 6 months and 1 year following discharge
Reporting Status: Not Posted

5. Secondary Outcome: First Bowel Movement
Description: Time to first bowel movement (# of days)
Time Frame: In-patient hospital stay, average 4-5 days
Reporting Status: Not Posted

6. Secondary Outcome: Anti-nausea Consumption
Description: Total in-hospital cumulative anti-nausea consumption
Time Frame: In-patient hospital stay, average 4-5 days
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Recovery
Description: Quality of Recovery (QOR) score (0-18)
Time Frame: In-patient hospital stay, first post operative 48 hours
Reporting Status: Not Posted

8. Secondary Outcome: Duration of Hospital Stay
Description: Duration of hospital stay (# of days)
Time Frame: In-patient hospital stay, average of 4-5 days
Reporting Status: Not Posted

9. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Postoperative nausea and vomiting (score of 0-3)
Time Frame: In Hospital postoperative measures, average 4-5 days
Reporting Status: Not Posted

10. Secondary Outcome: Sedation Level
Description: Sedation score in-patient
Time Frame: In Hospital postoperative measures, average 4-5 days
Reporting Status: Not Posted

11. Secondary Outcome: Pain Frequency and Intensity
Description: Short-form McGill Pain Questionnaire Score
Time Frame: Hospital discharge, average 4-5 days, 6 months and 1 year following discharge
Reporting Status: Not Posted

12. Secondary Outcome: Anxiety and Depression
Description: Hospital Anxiety and Depression Scale Score
Time Frame: Hospital discharge, average 4-5 days, 6 months and 1 year following discharge
Reporting Status: Not Posted

13. Secondary Outcome: Health Related Quality of Life
Description: Short-form health-related quality of life 36 Scores
Time Frame: Hospital discharge, average 4-5 days, 6 months and 1 year following discharge
Reporting Status: Not Posted

14. Secondary Outcome: Time to Ambulation
Description: Time to ambulation (# of days)
Time Frame: In-patient hospital stay, average 4-5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Isotonic Saline (Control Group) | Bupivacaine (Study Group)
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/49
Other Adverse Events (participants affected / at risk) | 2/44 | 3/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isotonic Saline (Control Group) (N=44) | Bupivacaine (Study Group) (N=49)
hematoma or revision of vessel anastomoses (Surgical and medical procedures) | 2 (2) | 3 (3) — Surgical evacuation of breast hematoma following breast reconstruction surgery

LIMITATIONS AND CAVEATS:
The study limitations include the difficulty in capturing data at all points postoperatively. The repeated measure pain scores at rest and with movement were not recorded for all patients (recorded for 75% at rest and 53% with movement).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No